CLINICAL TRIAL: NCT00849719
Title: Effects of Combination of Continuous Intravenous (IV) Infusion Plus Patient-Controlled Analgesia (PCA) of Morphine (MO) vs. IV-PCA MO on Postoperative Pain Control
Brief Title: Effects of a Combination of IV-PCA With Continuous IV Infusion of MO, Versus IV-PCA MO on Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Prof Avi Weinbrum, Director Post Anesthesia Care Unit, Tel Aviv Sourasky medical center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TASMC-08-AW-0400-CTIL
Record Dates: First submitted 2009-02-17; First posted 2009-02-24 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Post Operative Pain
Keywords: visual analog scale; patient controlled analgesia; post operative pain; rescue drug
MeSH Terms: conditions — Pain, Postoperative | interventions — Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients in this arm will recieve a combination of PCA MO (10 ug/kg/bolus, by request) and continuous infusion of MO (10 ug/kg/h), when visual analog scale (VAS) exeeds 5/10 boluses will be self-administered by the patient.
  Interventions: Drug: a combination of PCA MO and continuous infusion of MO
- 2 (Active Comparator): Patients in this arm will be administered with only boluses of 1.5 mg/bolus of MO, by request.
  Interventions: Drug: PCA MO only

INTERVENTIONS:
Drug: a combination of PCA MO and continuous infusion of MO — Patients in this arm will recieve a combination of PCA MO (10 ug/kg/bolus, by request) and continuous infusion of MO (10 ug/kg/h), when visual analog scale (VAS) exeeds 5/10 boluses will be self-administered by the patient. Rescue diclofenac 75 mg IM will be allowed once to help prompt start analgesia instead of opioid titration, and 6h later. No hourly dose limit will be set for the protocols.
  Other Names: PCA and infusion MO
  Arms: 1
Drug: PCA MO only — When visual analog scale [VAS] exeeds 5/10, and after the PACU drug-blinded attending physician had established that the patient is coherent and cooperative, a PCA system will be connected to the patient's IV line. The physician will start device, and deliver the first bolus. The subsequent drug boluses will be self-administered by the patient. Group 2 will be administered with only boluses of 1.5 mg/bolus of MO, by request. Rescue diclofenac 75 mg IM will be allowed once to help prompt start analgesia instead of opioid titration, and 6h later. No hourly dose limit will be set for the protocols.
  Other Names: PCA MO
  Arms: 2

SUMMARY:
After major surgery, such as abdominal or thoracic surgery, the majority of patients experience moderate to severe pain that may not be optimally controlled. Inadequate pain relief may lead to complications that can hinder rehabilitation and slow recovery. Morphine (MO) is the most commonly used opioid for the treatment of post-surgical pain (14). The preferred method of administration nowadays is intravenous patient-controlled analgesia (PCA). In contrast, Continuous infusion of intravenous morphine (CIVM) is seldom used in Post-Anesthesia Care Units (PACUs) for acute postoperative pain, due to concerns of cardio-respiratory deterioration, even though different studies have found this technique of administration effective and safe (in terms of opioid-related symptoms.As part of our efforts to improve postoperative pain management in the Tel Aviv Sourasky Medical Center's PACU, we wish to determine if combining CIVM with IV PCA will be superior over IV PCA only for the treatment of postoperative pain following major abdominal or thoracic surgery.Our hypothesis is that the continuous infusion, even if given at a relatively low dose, would enable the build-up of pharmacologically effective MO blood level, thus providing an overall better control of pain.

DETAILED DESCRIPTION:
Study objective To compare the efficacy of two MO administration-protocols: PCA MO (only) vs combination of continuous background infusion plus PCA MO (combined dosage) in patients after abdominal and thoracic surgery.

Methods Inclusion criteria The study will be conducted as a prospective, randomized, double blinded one, into which we will enroll patients aged 18-80 years undergoing major abdominal procedures (e.g. laparotomy, nephrectomy, gastrectomy, gastric bypass, pancreatectomy, splenectomy, and abdominal aortic aneurysm) or thoracic surgery (segmentectomy, lobectomy or pneumonectomy) in our institution during the years 2008-9.

Exclusion criteria We will exclude from the study patients with a history of drug or alcohol abuse, psychiatric disturbances, senile dementia, Alzheimer's disease, seizures or suicide risk, use of psychotropic drugs, pregnancy or nursing, hypersensitivity to MO, or to non steroidal anti-inflammatory drugs (NSAIDs) or their excipients, chronic or acute pain of any origin, respiratory failure or insufficiency, uncompensated or congestive heart or hepatic failure and those scheduled for an emergency or palliative procedure. We will also exclude patients using antidepressants, anticonvulsants or muscle relaxants, and patients using any monoamine oxidase inhibitor within 2 weeks of surgery.

Post enrollment dropouts Patients will be dropped from the study for one of the following reasons: need for immediate postoperative artificial ventilation lasting over 4 h, lack of coherence (<5/10) or constant sedation (>5/10 VAS), or combative behavior in the PACU, postoperative requirement for re-intervention and/or transfer to an intensive care unit (ICU). Other suitable patients will be recruited to replace the ones that were dropped.

Intra-study non-replaced dropouts will include protocol violation, patient's decision to withdraw or ineffective drug protocol (pain >5/10 VAS despite full and evidenced protocol implementation).

Intra-operative management Anesthetics and surgical management will be performed similarly in all patients. All patients will receive prophylactic antibiotics. All will be premedicated with oral 10 mg diazepam the night before surgery and 40-75 min preoperatively. After a sedative dose of IV midazolam (1.5-2 mg) and fentanyl (1.5 μg/kg), propofol (1-2 mg/kg) will be slowly injected IV until the patient losses consciousness. A non-depolarizing muscle relaxant will enable endotracheal intubation.

General anesthesia will be maintained according to institutional protocol, using nitrous oxide/oxygen 2/1 L/min enriched with isoflurane, aiming at delivering 1 MAC anesthesia. A non-depolarizing muscle relaxant and fentanyl will be continually infused or given by repeated portions to maintain muscle relaxation and analgesia, and hemodynamic and ventilatory stability. Cardiovascular and respiratory parameters will be monitored in the standard manner, and intraoperative fluid administration and blood replacement will follow common cardiovascular, renal and laboratory indices.

Towards the end of surgery, all drugs will be turned off and minimal doses of atropine and neostigmine will be administered to reverse muscle relaxation and obtain the return of normal spontaneous respiration. All patients will then be transferred to the PACU for observation.

Study design Consented postoperative patients will be randomly assigned to one of two groups (by using a closed-envelope technique): Group 1 will receive PCA bolus injections of MO, as practiced in our institution, whereas group 2 will receive both a basal (infusion) administration and PCA bolus injections. Dosage of the basal infusion and the PCA combination will be based on a preliminary dose-response pain control study and data obtained during a previous study, where the technique provided satisfactory reduction or even elimination of pain along with a tolerable level of side effects. For reasons of both safety and efficacy, we will maintain the doses of both basal (infusion) and demand (bolus) portions on a body weight basis.

Study phase and drug use Upon arrival in the PACU, each patient will be connected to an oxygen face-mask and a vital signs monitor. Upon the first complaint of moderate or severe rest pain (≥5/10 on a visual analog scale [VAS]), and after the PACU drug-blinded attending physician had established that the patient is coherent and cooperative, a PCA system will be connected to the patient's IV line. The physician will start device, and deliver the first bolus. The subsequent drug boluses will be self-administered by the patient. Group 1 patients will receive MO infusion (10 μg/kg/h) + MO bolus (10 μg/kg/bolus, by request), whereas group 2 will be administered with only boluses of 1.5 mg/bolus of MO. A 7 min lockout time after each bolus will prevent excessive dispensing of the drug. If needed, the physician could administer two extra boluses for optimal pain control within the first 15 min postoperatively. Rescue diclofenac 75 mg IM will be allowed once to help prompt start analgesia instead of opioid titration, and 6h later. No hourly dose limit will be set for the protocols.

All patients will be treated according to their designated study protocol for as long as they need; no use for 12 h after will prompt the patients to the standard pain care of the surgical department.

Patient assessment Outcome measurements will be assessed and documented every 15 min during the first 2 h of the study and then hourly, until POD3. Primary outcomes will include the demand/delivery ratio for MO and rescue drug (assessed by the hourly activation of the IV-PCA device, and the 12 h total drug consumption). Secondary outcomes will be: pain intensity (evaluated by both by the patients' self-rated pain, and via VAS by a blinded assessor), self-rated levels of sedation and satisfaction, time of dependence of the device and urinary catheter, time to discharge, and time until the patient sits, stand and leaves bed. Adverse effects that we will evaluate are: respiratory depression (respiratory rate, room air saturation, time to extubation in re-intubated patients); vomiting/nausea; allergic events, severe complications (e.g. morbidity).

The demographic data (age, gender, weight), background characteristics (pre-study heart and respiratory rates, SpO2, systolic and diastolic blood pressures), patients' American Society of Anesthesiologists (ASA) physical class, duration of surgery and intraoperative fentanyl usage will also be recorded; all will be analyzed at the end of the study.

Study hypothesis and benefits The present study aims at assessing whether the addition of MO infusion to the commonly used PCA, although both at a total dose that is inferior to that currently used in our institution, will provide better pain control compared to the commonly used technique. We believe that if this occurs, it will be safer for the patient and possibly allow earlier recovery, rehabilitation and home discharge.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing major abdominal procedures (e.g. laparotomy, nephrectomy, gastrectomy, gastric bypass, pancreatectomy, splenectomy, and abdominal aortic aneurysm) or thoracic surgery (segmentectomy, lobectomy or pneumonectomy) in our institution during the years 2008-9.

Exclusion Criteria:

* patients with a history of drug or alcohol abuse, psychiatric disturbances, senile dementia, Alzheimer's disease, seizures or suicide risk, use of psychotropic drugs, pregnancy or nursing, hypersensitivity to MO, or to non steroidal anti-inflammatory drugs (NSAIDs) or their excipients, chronic or acute pain of any origin, respiratory failure or insufficiency, uncompensated or congestive heart or hepatic failure and those scheduled for an emergency or palliative procedure.
* we will also exclude patients using antidepressants, anticonvulsants or muscle relaxants, and patients using any monoamine oxidase inhibitor within 2 weeks of surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-04 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
demand/delivery ratio for MO and rescue drug | hourly and 12 h total drug consumption

SECONDARY OUTCOMES:
pain intensity | hourly

CONTACTS AND LOCATIONS:
Overall Officials: Avi Weinbrum, MD, Study Chair — Director Post Anesthesia Care Unit, TASMC
Locations (1):
- Tel Aviv Sourasky medical center, Tel Aviv, Israel

REFERENCES:
- [Background] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949